CLINICAL TRIAL: NCT02235844
Title: Allogeneic Transplantation of Human Umbilical Cord Mesenchymal Stem Cells (UC-MSC) for a Single Male Patient With Duchenne Muscular Dystrophy (DMD)
Brief Title: Allogeneic Human Umbilical Cord Mesenchymal Stem Cells for a Single Male Patient With Duchenne Muscular Dystrophy (DMD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergy and Asthma Consultants, Wichita, Kansas (Other)
Collaborators: Aidan Foundation (Unknown); Neil H. Riordan PhD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND 16026 DMD Single Patient
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Duchenne's Muscular Dystrophy
Keywords: Mesenchymal; Stem Cells; Umbilical Cord; Duchenne's; Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Mesenchymal Stem Cells (Experimental): Umbilical Cord Mesenchymal Stem Cells
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Umbilical Cord Mesenchymal Stem Cells

SUMMARY:
This research study is designed to evaluate the effects of human umbilical cord mesenchymal stem cells (UC-MSCs), on Duchenne's muscular dystrophy (DMD). The potential muscle regenerative and anti-inflammatory properties of UC MSCs position them as a possible treatment option for DMD. Both of these properties could lead to potential benefits for a DMD patient.

ELIGIBILITY:
Inclusion Criteria:

* Duchenne's Muscular Dystrophy

Exclusion Criteria:

* None

Ages: 28 Years to 31 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 3 months after final treatment
  No occurrence of adverse events

SECONDARY OUTCOMES:
Change from baseline of weight | 3 months after final treatment
Change of muscle diameter (circumferential measurements) from baseline | 3 months after final treatment
Change from baseline of Pulmonary Maximum Expiratory Pressure | 3 months after final treatment
Change from baseline of Pulmonary Forced Vital Capacity | 3 months after final treatment
Maximum Change from baseline of Predicted Inspiratory Pressure % | 3 months after final treatment
Change from baseline of Predicted Maximum Expiratory Pressure % | 3 months after final treatment
Change from baseline of Predicted Forced Vital Capacity % | 3 months after final treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maurice HV Strickland, MD, Principal Investigator — Allergy and Asthma Consultants of Wichita, KS
Locations (1):
- Asthma and Allergy Consultants, Wichita, Kansas, United States